CLINICAL TRIAL: NCT04199715
Title: Immunologic Efficacy of Heplisav B Vaccine in Patients Undergoing Treatment With Immunosuppressive Medications
Brief Title: Safety and Efficacy of a Hepatitis B Vaccine in Immunosuppressed Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IND 18850
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Hep B; Vaccine; Immunosuppression; HBV
MeSH Terms: conditions — Hepatitis B | interventions — Heplisav-B

STUDY DESIGN:
Intervention Model Description: A total of 18 patients will be entered into the study including 3 evenly sized groups of 6 as follows:
  * Group A patients on tumor necrosis factor alpha or interleukin inhibitor therapy for underlying chronic inflammatory disorders
  * Group B patients on chemotherapy for solid organ malignancy
  * Group C patients are either recipients of livers from anti-HBc positive donors or are patients transplanted for chronic hepatitis B infection without recurrent hepatitis B at the time of enrollment
Masking Description: N/A. Investigator and patient will know that the patient received the Heplisav-B vaccine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Heplisav-B Vaccine Recipient (Experimental): There will be a single group of 18 immune compromised patients who will receive the Heplisav-B vaccine.
  Interventions: Biological: Heplisav-B

INTERVENTIONS:
Biological: Heplisav-B — This is an FDA-approved vaccine for Hepatitis B that is made by Dynavax Technologies.

SUMMARY:
This is a preliminary trial of a Hepatitis B vaccine (Heplisav-B) in medically immunosuppressed patients. The purpose of this study is to test the ability of Heplisav-B to produce high levels of antibody that neutralize the virus and prevent hepatitis B from coming back. Another important purpose is to test the safety of this vaccine in patients taking immune suppressive medicines.

DETAILED DESCRIPTION:
This is an open label exploratory study of the immunologic efficacy and safety of an FDA-approved Hepatitis B vaccine called Heplisav-B. It will be used in patients treated with long term immunosuppressive drug therapy. The patients will be given two doses of Heplisav-B, the first delivered at the baseline visit and the second at week 4. Antibody levels against the Hepatitis B virus will be measured at baseline and at weeks 4, 8, 12, 24 and 60. The proportion of those patients with protective antibody levels will be compared with non-immune compromised patients receiving the same dosing schedule. Patients who fail to demonstrate protective levels of antibodies at week 8 will be given a third booster dose at week 12, and all patients will be followed to week 60.

This research is being done because current alternative hepatitis B vaccines produce lower levels of antibody to hepatitis B, and the level of antibody can be important in the prevention of the virus coming back. However, administration of Heplisav-B has been associated with higher levels of protective antibody in healthy individuals, people with diabetes, and people with kidney disease. It is hoped that the same beneficial effect of higher antibody level will also occur in patients who take an immune suppressing medicine to treat underlying inflammatory disorder (either arthritis, colitis, or chronic skin inflammation), chemotherapy for cancer, or anti-rejection therapy for liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older and agree to adhere to study requirements
* Must be willing to provide informed consent
* Serologic profile consistent with resolved hepatitis B (HBsAg negative but anti-HBc positive)
* Must meet one of the following requirements: Recipient of anti-HBc positive liver (Group C), Chronic inflammatory disease requiring TNF or interleukin inhibitor therapy (Group A), Solid organ malignancy that requires systemic cancer chemotherapy (Group B), or Post liver transplant for chronic HBV infection (Group C).
* Recipient of immunosuppressive drug medication as described above

Exclusion Criteria:

* HBsAg positivity
* Anti-HBs level > 20 mIU/mL at baseline
* HIV infection
* HCV infection
* Prior hepatitis B vaccination
* Received hepatitis B immune globulin during the past 4 months
* Hematologic malignancy
* Hepatocellular carcinoma
* Active alcohol use > 20 grams daily
* Unstable underlying inflammatory disorder
* Pregnancy or breast feeding
* History of severe depression or other severe psychiatric disorder
* Received liver transplant < 3 years earlier
* Transplant rejection within the past year
* Unstable or poorly responsive inflammatory disorders
* Patients who have an unreasonable risk of complications
* Anticipated life expectancy less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Safety of Heplisav-B Vaccine in Immunosuppressed Patients | 60 weeks
  Patients will be followed for 60 weeks to capture adverse events. Safety will be determined by the proportion of patients with unsolicited adverse events after vaccine administration, the proportion of patients with serious adverse events, the proportion of patients with medically attended adverse events, the proportion of patients with potentially immune-mediated medical conditions, and the proportion of patients who need an increase in immune suppressive medication.
Immunologic Efficacy of Heplisav-B Vaccine in Immunosuppressed Patients | 60 weeks
  Efficacy will be determined by the proportion of patients who respond with seroprotective levels (> 10 mIU/ml) of anti-HBs at each study interval and the proportion of patients with anti-HBs titers > 100 mIU/ml at each study interval.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Perrillo, MD, FAASLD, Principal Investigator — Baylor Scott & White Research Institute
Locations (1):
- Baylor Scott & White Research Institute, Dallas, Texas, United States

REFERENCES:
- [Background] Schillie S, Vellozzi C, Reingold A, Harris A, Haber P, Ward JW, Nelson NP. Prevention of Hepatitis B Virus Infection in the United States: Recommendations of the Advisory Committee on Immunization Practices. MMWR Recomm Rep. 2018 Jan 12;67(1):1-31. doi: 10.15585/mmwr.rr6701a1. PMID 29939980
- [Background] Paul S, Dickstein A, Saxena A, Terrin N, Viveiros K, Balk EM, Wong JB. Role of surface antibody in hepatitis B reactivation in patients with resolved infection and hematologic malignancy: A meta-analysis. Hepatology. 2017 Aug;66(2):379-388. doi: 10.1002/hep.29082. Epub 2017 Jun 22. PMID 28128861
- [Background] Splawn LM, Bailey CA, Medina JP, Cho JC. Heplisav-B vaccination for the prevention of hepatitis B virus infection in adults in the United States. Drugs Today (Barc). 2018 Jul;54(7):399-405. doi: 10.1358/dot.2018.54.7.2833984. PMID 30090877
- [Derived] Perrillo R, Garrido LF, Ma TW, Rahimi R, Lilly B. Vaccination with HepB-CpG vaccine in individuals undergoing immune suppressive drug therapy. Vaccine. 2023 Jul 12;41(31):4457-4461. doi: 10.1016/j.vaccine.2023.06.041. Epub 2023 Jun 21. PMID 37353450

DOCUMENTS (1):
  • Study Protocol (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT04199715/Prot_000.pdf